CLINICAL TRIAL: NCT03889444
Title: Drug Utilization Study in Patients Receiving Ozurdex™ (Dexamethasone Intravitreal Implant) 0.7 mg Injections for Visual Impairment Due to Diabetic Macular Edema (DME)
Brief Title: Chart Review: Drug Utilization Study in Participants Who Received Ozurdex™ (Dexamethasone Intravitreal Implant) 0.7 mg Injections for Visual Impairment Due to Diabetic Macular Edema (DME)
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: CMO-MA-EYE-0564
Record Dates: First submitted 2019-03-07; First posted 2019-03-26 (Actual); Results first posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-05

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OZURDEX®: Participants with diabetic macular edema prescribed dexamethasone intravitreal implant, 0.7 mg (OZURDEX®) as per routine clinical practice.
  Interventions: Drug: Dexamethasone intravitreal implant

INTERVENTIONS:
Drug: Dexamethasone intravitreal implant — Dexamethasone intravitreal implant 0.7 mg injection, as per routine clinical practice.
  Other Names: OZURDEX®

SUMMARY:
A retrospective, non-interventional, observational, multi-center, drug utilization study to be conducted in adult participants with visual impairment due to DME treated with Ozurdex implants in Germany and Switzerland from 1 January 2015 to 1 September 2017.

ELIGIBILITY:
Inclusion Criteria:

* Participant received at least two Ozurdex® implants in the study eye to treat visual impairment due to DME
* First Ozurdex® implant injection occurred after 1 January 2015
* Participant was followed-up at the site for at least 12 months after the first Ozurdex® implant in the study eye

Exclusion Criteria:

- Participant received Ozurdex® implants as part or during a clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From a public health and market access perspective, the present study population constitutes a broader real-world participant population than that reflected in clinical trials. The present study design does not make any conclusions on causal relationships, but can rather explore real-world Ozurdex® drug utilization patterns, effectiveness and safety. It is expected that the results from this study may be generalizable to the overall population presenting with DME and treated with Ozurdex® in Germany and Switzerland. Participants may contribute at most one eye into the study. If both eyes meet the inclusion criteria, the eye that received the most Ozurdex® injections will be chosen as the study eye.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paramjit Singh, Study Director — Allergan
Locations (1):
- Clinical Trials Registry Team, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance. — http://AllerganClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OZURDEX®
Started | 141
Completed | 141
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis Population included all selected participants for whom an electronic case report form (eCRF) has been completed and who met selection criteria.
Arm/Group | OZURDEX®
Number analyzed (Participants) | 141
Age, Continuous [Mean (Full Range); unit: years] | 65.7 [31 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 84
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of OZURDEX® Implant Reinjections in the Study Eye
Description: Study eye was defined as the eye that received the most OZURDEX® injections.
Time Frame: Up to 44 months
Population: Analysis Population included all selected participants for whom an eCRF has been completed and who met selection criteria.
Measure: Mean (Standard Deviation); unit: number of injections
Arm/Group | OZURDEX®
Number analyzed (Participants) | 141
number of injections | 3.0 (1.9)

2. Primary Outcome: Time to OZURDEX® Reinjection
Description: The time to reinjection is defined as the time in months from the date of one OZURDEX® injection to the subsequent OZURDEX® injection.
Time Frame: Up to 44 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: months
Arm/Group | OZURDEX®
Number analyzed (Participants) | 141
months | 5.7 (4.2)

3. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA) From the Last Assessment Prior to Each OZURDEX® Implant Injection to 7-12 Weeks Following Each OZURDEX® Implant Injection
Description: BCVA is measured in the study eye (defined as the eye that received the most OZURDEX® injections) following each injection of OZURDEX® using a special eye chart and is reported as number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision. The higher the number of letters read correctly, the better the vision. A positive number indicates improvement. Change data are reported for each injection relative to the assessment immediately prior to the injection to 7 to 12 weeks following that injection.
Time Frame: Last assessment prior to each OZURDEX® injection, 7 to 12 weeks following each injection
Population: Analysis Population included all selected participants for whom an eCRF has been completed and who met selection criteria. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | OZURDEX®
Number analyzed (Participants) | 141
letters
  Before Injection 1 to 7-12 weeks After Injection 1: number analyzed (Participants) | 77
  Before Injection 1 to 7-12 weeks After Injection 1 | 3.4 (13.7)
  Reinjection 1 to 7-12 weeks After Reinjection 1: number analyzed (Participants) | 30
  Reinjection 1 to 7-12 weeks After Reinjection 1 | 1.2 (12.4)
  Reinjection 2 to 7-12 weeks After Reinjection 2: number analyzed (Participants) | 21
  Reinjection 2 to 7-12 weeks After Reinjection 2 | 0.5 (5.8)
  Reinjection 3 to 7-12 weeks After Reinjection 3: number analyzed (Participants) | 10
  Reinjection 3 to 7-12 weeks After Reinjection 3 | 3.2 (8.0)
  Reinjection 4 to 7-12 weeks After Reinjection 4: number analyzed (Participants) | 6
  Reinjection 4 to 7-12 weeks After Reinjection 4 | 3.0 (4.7)
  Reinjection 5 to 7-12 weeks After Reinjection 5: number analyzed (Participants) | 4
  Reinjection 5 to 7-12 weeks After Reinjection 5 | 0.1 (4.7)
  Reinjection 6 to 7-12 weeks After Reinjection 6: number analyzed (Participants) | 3
  Reinjection 6 to 7-12 weeks After Reinjection 6 | -0.3 (0.6)
  Reinjection 7 to 7-12 weeks After Reinjection 7: number analyzed (Participants) | 1
  Reinjection 7 to 7-12 weeks After Reinjection 7 | 0.0 (NA) — Standard deviation (SD) was not estimable for one participant.
  Reinjection 8 to 7-12 weeks After Reinjection 8: number analyzed (Participants) | 2
  Reinjection 8 to 7-12 weeks After Reinjection 8 | 6.3 (8.8)
  Reinjection 9 to 7-12 weeks After Reinjection 9: number analyzed (Participants) | 2
  Reinjection 9 to 7-12 weeks After Reinjection 9 | -0.5 (0.7)
  Reinjection 10 to 7-12 weeks After Reinjection 10: number analyzed (Participants) | 2
  Reinjection 10 to 7-12 weeks After Reinjection 10 | 0.0 (0.0)

4. Secondary Outcome: Change From Baseline in BCVA From the Last Assessment Prior to the First OZURDEX® Implant Injection to 7-12 Weeks Following Each OZURDEX® Implant Injection
Description: BCVA is measured in the study eye (defined as the eye that received the most OZURDEX® injections) following each injection of OZURDEX® using a special eye chart and is reported as number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision. The higher the number of letters read correctly, the better the vision. A positive change from baseline indicates improvement. Change data are reported for each injection relative to the assessment prior the first injection to 7 to 12 weeks following each injection.
Time Frame: Baseline (Last assessment prior to the first OZURDEX® injection), 7 to 12 weeks following each injection
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | OZURDEX®
Number analyzed (Participants) | 141
letters
  Baseline to 7-12 weeks After Injection 1: number analyzed (Participants) | 77
  Baseline to 7-12 weeks After Injection 1 | 3.4 (13.7)
  Baseline to 7-12 weeks After Reinjection 1: number analyzed (Participants) | 71
  Baseline to 7-12 weeks After Reinjection 1 | 3.7 (10.0)
  Baseline to 7-12 weeks After Reinjection 2: number analyzed (Participants) | 42
  Baseline to 7-12 weeks After Reinjection 2 | 3.2 (10.9)
  Baseline to 7-12 weeks After Reinjection 3: number analyzed (Participants) | 32
  Baseline to 7-12 weeks After Reinjection 3 | -1.4 (12.5)
  Baseline to 7-12 weeks After Reinjection 4: number analyzed (Participants) | 20
  Baseline to 7-12 weeks After Reinjection 4 | 0.5 (18.6)
  Baseline to 7-12 weeks After Reinjection 5: number analyzed (Participants) | 13
  Baseline to 7-12 weeks After Reinjection 5 | 3.5 (15.4)
  Baseline to 7-12 weeks After Reinjection 6: number analyzed (Participants) | 7
  Baseline to 7-12 weeks After Reinjection 6 | 5.1 (8.2)
  Baseline to 7-12 weeks After Reinjection 7: number analyzed (Participants) | 3
  Baseline to 7-12 weeks After Reinjection 7 | 0.0 (0.0)
  Baseline to 7-12 weeks After Reinjection 8: number analyzed (Participants) | 3
  Baseline to 7-12 weeks After Reinjection 8 | -0.8 (3.8)
  Baseline to 7-12 weeks After Reinjection 9: number analyzed (Participants) | 3
  Baseline to 7-12 weeks After Reinjection 9 | -3.7 (3.2)
  Baseline to 7-12 weeks After Reinjection 10: number analyzed (Participants) | 3
  Baseline to 7-12 weeks After Reinjection 10 | -0.3 (4.5)

5. Secondary Outcome: Change in Central Retinal Thickness (CRT) by Optical Coherence Tomography (OCT) From the Last Assessment Prior to Each OZURDEX® Implant Injection to 7-12 Weeks Following Each OZURDEX® Implant Injection
Description: OCT is measured in the study eye (defined as the eye that received the most OZURDEX® injections) prior to and following each injection of OZURDEX®. OCT is a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina to assess retinal thickness. A negative change indicates an improvement. Change data are reported for each injection relative to the assessment immediately prior to the injection to 7 to 12 weeks following that injection.
Time Frame: Last assessment prior to each OZURDEX® injection, 7 to 12 weeks following each injection
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: micrometer (μm)
Arm/Group | OZURDEX®
Number analyzed (Participants) | 141
micrometer (μm)
  Before Injection 1 to 7-12 weeks After Injection 1: number analyzed (Participants) | 69
  Before Injection 1 to 7-12 weeks After Injection 1 | -88.3 (100.2)
  Reinjection 1 to 7-12 weeks After Reinjection 1: number analyzed (Participants) | 22
  Reinjection 1 to 7-12 weeks After Reinjection 1 | -63.9 (79.6)
  Reinjection 2 to 7-12 weeks After Reinjection 2: number analyzed (Participants) | 15
  Reinjection 2 to 7-12 weeks After Reinjection 2 | -70.4 (96.4)
  Reinjection 3 to 7-12 weeks After Reinjection 3: number analyzed (Participants) | 10
  Reinjection 3 to 7-12 weeks After Reinjection 3 | -51.6 (54.4)
  Reinjection 4 to 7-12 weeks After Reinjection 4: number analyzed (Participants) | 3
  Reinjection 4 to 7-12 weeks After Reinjection 4 | -84.0 (94.4)
  Reinjection 5 to 7-12 weeks After Reinjection 5: number analyzed (Participants) | 4
  Reinjection 5 to 7-12 weeks After Reinjection 5 | -60.6 (44.2)
  Reinjection 6 to 7-12 weeks After Reinjection 6: number analyzed (Participants) | 3
  Reinjection 6 to 7-12 weeks After Reinjection 6 | -68.3 (93.9)
  Reinjection 7 to 7-12 weeks After Reinjection 7: number analyzed (Participants) | 1
  Reinjection 7 to 7-12 weeks After Reinjection 7 | -3.0 (NA) — SD was not estimable for one participant.
  Reinjection 8 to 7-12 weeks After Reinjection 8: number analyzed (Participants) | 1
  Reinjection 8 to 7-12 weeks After Reinjection 8 | -70.0 (NA) — SD was not estimable for one participant.
  Reinjection 9 to 7-12 weeks After Reinjection 9: number analyzed (Participants) | 2
  Reinjection 9 to 7-12 weeks After Reinjection 9 | -55.5 (4.9)
  Reinjection 10 to 7-12 weeks After Reinjection 10: number analyzed (Participants) | 2
  Reinjection 10 to 7-12 weeks After Reinjection 10 | -15.0 (2.8)

6. Secondary Outcome: Change From Baseline in CRT by OCT From the Last Assessment Prior to the First OZURDEX® Implant Injection to 7-12 Weeks Following Each OZURDEX® Implant Injection
Description: OCT is measured at Baseline and following each injection of OZURDEX® in the study eye (defined as the eye that received the most OZURDEX® injections . OCT is a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina to assess retinal thickness. A negative change indicates an improvement. Change data are reported for each injection relative to the assessment prior the first injection to 7 to 12 weeks following each injection.
Time Frame: Baseline (Last assessment prior to the first OZURDEX® injection), 7 to 12 weeks following each injection
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | OZURDEX®
Number analyzed (Participants) | 141
μm
  Baseline to 7-12 weeks After Injection 1: number analyzed (Participants) | 69
  Baseline to 7-12 weeks After Injection 1 | -88.3 (100.2)
  Baseline to 7-12 weeks After Reinjection 1: number analyzed (Participants) | 52
  Baseline to 7-12 weeks After Reinjection 1 | -81.6 (97.5)
  Baseline to 7-12 weeks After Reinjection 2: number analyzed (Participants) | 36
  Baseline to 7-12 weeks After Reinjection 2 | -102.4 (117.6)
  Baseline to 7-12 weeks After Reinjection 3: number analyzed (Participants) | 26
  Baseline to 7-12 weeks After Reinjection 3 | -124.1 (165.1)
  Baseline to 7-12 weeks After Reinjection 4: number analyzed (Participants) | 16
  Baseline to 7-12 weeks After Reinjection 4 | -115.7 (135.6)
  Baseline to 7-12 weeks After Reinjection 5: number analyzed (Participants) | 11
  Baseline to 7-12 weeks After Reinjection 5 | -147.7 (152.6)
  Baseline to 7-12 weeks After Reinjection 6: number analyzed (Participants) | 7
  Baseline to 7-12 weeks After Reinjection 6 | -167.3 (244.4)
  Baseline to 7-12 weeks After Reinjection 7: number analyzed (Participants) | 3
  Baseline to 7-12 weeks After Reinjection 7 | -35.3 (29.0)
  Baseline to 7-12 weeks After Reinjection 8: number analyzed (Participants) | 2
  Baseline to 7-12 weeks After Reinjection 8 | -22.5 (6.4)
  Baseline to 7-12 weeks After Reinjection 9: number analyzed (Participants) | 3
  Baseline to 7-12 weeks After Reinjection 9 | -19.3 (91.6)
  Baseline to 7-12 weeks After Reinjection 10: number analyzed (Participants) | 3
  Baseline to 7-12 weeks After Reinjection 10 | -42.3 (62.1)

7. Secondary Outcome: Percentage of Participants Who Experienced At Least One Adverse Events of Special Interest (AESIs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the drug. The adverse events of special interest include: Glaucoma, defined as damage to the optic nerve with progressive vision loss, Intraocular hypertension, defined as intra-ocular pressure (IOP) without meeting the criteria for glaucoma, Hypotony, defined as low IOP ≤5 mmHg, Cataract or lens opacities, Ocular bleeding or hemorrhage, Retinal detachment, tear or hole, Vitreous detachment, Infection vs. Non-infection related Ocular inflammation, Significant vitreous loss, Mechanical failure of device and implant misplacement, Implant dislocation.
Time Frame: Up to 44 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | OZURDEX®
Number analyzed (Participants) | 141
percentage of participants | 18.4

ADVERSE EVENTS:
Time Frame: Up to 44 months
Description: Only adverse events of special interest were collected during the study.
Arm/Group | OZURDEX®
All-Cause Mortality (participants affected / at risk) | 0/141
Serious Adverse Events (participants affected / at risk) | 0/141
Other Adverse Events (participants affected / at risk) | 16/141
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OZURDEX® (N=141)
Intraocular hypertension (Eye disorders) | 9
Cataract or lens opacities (Eye disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/44/NCT03889444/SAP_000.pdf
  • Study Protocol (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/44/NCT03889444/Prot_001.pdf